CLINICAL TRIAL: NCT07399379
Title: Implementation of an Augmented Reality System to Complement Discharge Information in Hospitalized Cardiology Patients
Brief Title: Augmented Reality as Discharge Information for Hospitalized Cardiology Patients
Acronym: RACAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEIm 23/44; SEC/FEC-INV-CLI 23/12 (Other Grant/Funding Number: Spanish Society of Cardiology)
Record Dates: First submitted 2026-01-13; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Myocardial Infarction (MI); Pacemaker Implantation; Heart Failure; Atrial Fibrillation (AF)
Keywords: Augmented reality; Acute Coronary Syndrome; Heart Failure; Pacemaker; PREM; Atrial Fibrillation
MeSH Terms: conditions — Myocardial Infarction; Heart Failure; Atrial Fibrillation; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): This group receives the usual medical discharge report plus an information card with a drawing and a QR code that gives access to an augmented reality application explaining their disease.
  Interventions: Device: Augmented reality app
- Control group (No Intervention): This group receives the usual medical discharge report.

INTERVENTIONS:
Device: Augmented reality app — The card provided in addition to the usual medical discharge report is designed with a simple drawing that identifies each condition and a QR code.
  This code can be scanned from any mobile device using the device's camera. Once scanned, a 3D model of a heart or a stent (depending on the condition) appears on the device, showing movement, vibration, and sound as an example of augmented reality.
  The user can also access simple options through three buttons:
  1. Video recorded by a cardiology professional: a brief and easy-to-understand explanation of the patient's condition, lasting approximately 2-3 minutes, provided by a hospital cardiology professional.
  2. Treatment recommendations: a drop-down section with a table of discharge recommendations for the patient's condition, including lifestyle and dietary advice.
  3. Warning signs: situations that the patient should pay attention to and seek medical advice if they occur.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to find out whether a simple augmented reality tool provided at hospital discharge can improve patients' understanding of their care, adherence to treatment, and health outcomes, compared with the usual discharge information.

This study includes adult patients who are admitted to a cardiology department because of:

* Ischaemic heart disease
* Atrial fibrillation
* Heart failure
* Or who need a pacemaker implantation

The main questions this study aims to answer are:

* Does providing augmented reality information at discharge improve patients' perceived quality of care?
* Does it improve patients' adherence to their prescribed treatment?
* Does it reduce major cardiovascular events such as hospital readmission, heart attack, stroke, or cardiovascular death?

Researchers will compare two groups of participants:

* A control group, who will receive the usual medical discharge report.
* An intervention group, who will receive the usual medical discharge report plus an information card with a drawing and a QR code that gives access to an augmented reality application.

Participants will:

* Receive their discharge information according to the group they are assigned to.
* Use the augmented reality application if they are in the intervention group.
* Be followed over time to assess treatment adherence, patient experience, and cardiovascular events.

This is a low-intervention, randomized, single-centre clinical trial conducted in Getafe, Madrid, Spain. Participation in this study does not involve taking any additional medication.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have access to a mobile device (such as a smartphone or tablet).
* Participants must have been admitted to the Cardiology Department of Getafe University Hospital for ischemic heart disease, heart failure, atrial fibrillation, or pacemaker implantation.

Exclusion Criteria:

* No access to a mobile device.
* Untreated visual or hearing impairments that prevent viewing or understanding the videos.
* Inability to understand Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
PRIMARY OUTCOME: PREM and treatment adherence at one and six months | Follow up at one and six months from enrollment
  To assess PREM (Patient-Reported Experience Measures) in the intervention group and in the control group at discharge and at follow-up.

SECONDARY OUTCOMES:
MACE at one and six months | From enrollment at one and six months
  Data on major adverse cardiovascular events (MACE) will also be collected at one and six months from discharge in both groups. MACE include heart attack, stroke, cardiovascular-related hospital readmission, and cardiovascular death.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Getafe, Getafe, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared because the dataset contains sensitive patient health information, including medical history and follow-up outcomes. Sharing these data could risk patient confidentiality. All data will be handled according to current data protection regulations and only anonymized, aggregated results will be made publicly available.

REFERENCES:
- [Background] Davies F. Perceived usefulness, perceived ease of use, and user acceptance of information technology. MIS Quarterly. 1989; 13: 319-40.
- [Background] Labanas V, Loukas C, Smailis N, et al. A novel augmented reality simulator for skills assessment in minimal invasive surgery. Surg Endosc. 2015; 29: 2224-34.
- [Background] Kang X, Azizian M, Wilson E, et al. Stereoscopic augmented reality for laparoscopic surgery. Surg Endosc. 2014; 28: 2227-35.
- [Background] Barroso Osuna, J., & Cabero Almenara, J. (2016). Evaluación de objetos de aprendizaje en Realidad Aumentada: estudio piloto en el grado de Medicina. Enseñanza & Teaching: Revista Interuniversitaria De Didáctica, 34(2), 149-67. https://doi.org/10.14201/et2016342149167.
- [Background] Almenara, J.C., Osuna, J.B., Puente, Á.P., et al. Realidad Aumentada para aumentar la formación en la enseñanza de la Medicina. Educ. Medica. Super. 2018; 32 (4): 1-14.